CLINICAL TRIAL: NCT04902963
Title: What is the Tympanic Membrane Healing Time After Insertion of a Gelfoam PE Tube?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skovlund Medical Products, LLC (Other)
Responsible Party: Principal Investigator, Sandra Skovlund, Primary Investigator, Skovlund Medical Products, LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 04053-10-C
Record Dates: First submitted 2021-04-01; First posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Eustachian Tube Dysfunction; Sudden Hearing Loss; Meniere Disease
MeSH Terms: conditions — Hearing Loss, Sudden; Meniere Disease

STUDY DESIGN:
Intervention Model Description: 14 patients underwent placement of a novel absorbable ventilation tube to test utility of this prototype device and monitor resorption over a period of weeks. 14 participants were approved for this study of feasibility to allow for patients who did not follow up per the study protocol.
Masking Description: 2 examiners used otomicroscopy to document the function of the ear tube by documenting the number of weeks the lumen remained patent and the number of weeks until the device was fully resorbed. All examiners documented results independent of the other examiner.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meeting indication for short term ventilation tube placement (Experimental): Adult patients meeting standard criteria for short-term ventilation tube placement were offered placement of a bioabsorbable ear tube in place of a durable ear tube that would later be removed.
  Interventions: Device: PE tube

INTERVENTIONS:
Device: PE tube — Gelatin mixed with antibiotic and steroid ear drop to create a rigid device that maintains a lumen, acting as an intermediate-duration bioabsorbable ear tube.

SUMMARY:
Pilot study done to evaluate the breakdown and and potential utility of a bioabsorbable ventilation ear tube made with gelatin.

DETAILED DESCRIPTION:
Institutional Review Board- Park Nicollet Institute approval was granted 3/2011 for 15 patients to be enrolled in pilot study of use of a bioabsorbable ventilation ear (PE) tube. IRB stated compliance with FDA as defined in 21 CFR, Part 56 and with regulations of DHHS. Federal assurance number FWA00000914. Prior to commencing this study, IRB approval was obtained and each participating clinician completed the NIH training for "Protecting Human Research Participants".

14 patients (15 ears) were enrolled in this study and were examined by 2 independent examiners at approximately 3, 6 and 12 week follow-ups. Lumen patency and time to complete resorption were documented by each examiner. There were no adverse reactions. This pilot study suggests that there is utility for a bioabsorbable ear tube made from gelatin material, as the device was found to break down over the expected time frame and remained functional long enough to have clinical utility.

ELIGIBILITY:
Inclusion Criteria:

* meeting indications for placement of a short or intermediate-duration ventilation ear tube (PE tube)

Exclusion Criteria:

* none

Ages: 26 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-03-15 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Number of weeks that ventilation tube lumen is patent. | 0-3 months
  Primary outcome was presence of a lumen, reflecting a functional device.

SECONDARY OUTCOMES:
Number of weeks until ventilation tube is fully resorbed. | 0-3 months
  Gelatin has been used in this site as packing material and has been shown to resorb over a period of several weeks. Full resorption of this device is expected.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Walker, Study Director — Park Nicollet Institute, IRB Administrator